CLINICAL TRIAL: NCT00000876
Title: Phase I/II Trial of CD4-IgG2 in HIV-Infected Children
Brief Title: Safety and Effectiveness of CD4-IgG2 in HIV-Positive Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PACTG 351; 10699 (Registry Identifier: DAIDS ES Registry Number); ACTG 351
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Antiviral Agents; CD4-IgG(2); PRO 542
MeSH Terms: conditions — HIV Infections | interventions — CD4-IgG(2)

INTERVENTIONS:
Drug: CD4-IgG2

SUMMARY:
CD4-IgG2 is a special man-made protein that was built to block the entrance of HIV into CD4 cells (cells of the immune system that fight infection). The purpose of this study is to see if giving CD4-IgG2 to HIV-infected children is safe and effective.

HIV attaches to CD4 cells and enters them. Inside, HIV makes copies of itself that will help the virus invade the body. CD4 cells are killed or disabled during this process of HIV replication. Decreases in CD4 cells lead to a weakened immune system. When CD4 cell counts become very low, the body is unable to defend itself, and HIV infection develops into AIDS. The protein used in this study, CD4-IgG2, may be able to attach to HIV and inactivate it so that it cannot enter CD4 cells. This is an early study to examine CD4-IgG2 as a possible treatment for HIV in children.

DETAILED DESCRIPTION:
Since CD4 is the high-affinity receptor for HIV-1, molecules such as CD4-IgG2, which incorporate the gp120 binding region of CD4, have the potential to bind and neutralize all strains of the virus. [AS PER AMENDMENT 4/25/00: Study results have demonstrated that the product is safe in children, well tolerated, and may have antiviral properties. With these encouraging results in hand, an extra cohort has been added using twice the dose of rCD4-IgG2 as in Cohort I.]

The study is conducted in two parts. In Part 1 patients receive a single dose of CD4-IgG2 intravenously at 1 of 4 dose levels. A minimum of 3 patients are treated at a given dose level. If none of these 3 patients experience Grade 3 or 4 toxicity, patients are escalated to the next dose level. If any of these 3 patients have life-threatening toxicities or if more than 1 of these 3 patients experience non-life-threatening Grade 3 or 4 toxicities, escalation stops and the prior dose (if any) is considered the maximum tolerated dose (MTD). If 1 of these 3 patients experiences non-life-threatening Grade 3 or 4 toxicities, 3 additional patients are treated at this dose level. If 1 or more of these 3 additional patients has Grade 3 or 4 toxicity, escalation stops. If none of these 3 additional patients has Grade 3 or 4 toxicity, patients are escalated to the next dose level.

Part 2 provides additional data on the safety, toxicity and pharmacokinetics of CD4-IgG2 when given in multiple doses. Patients receive the highest safe dose (MTD) as established in Part 1. Treatment is given intravenously once weekly at Weeks 0, 1, 2, and 3. If insufficient activity is seen at this dose level, 6 additional patients will be enrolled at a higher dose level. Patients who participate in Part 1 may enroll in Part 2 provided they are followed for at least 3 months and meet inclusion criteria for Part 2. If any patient experiences a life-threatening condition due to CD4-IgG2, the study will stop. [AS PER AMENDMENT 4/25/00: Cohort II receives twice the dose of Cohort I intravenously once weekly at Weeks 0, 1, 2 and 3. Pharmacokinetic samples are obtained at pre-dose and 1 hour after the doses are administered at Weeks 0, 1, and 2; and pre-dose, 1 hour, 24 hours, and Days 3, 7, and 14 after the dose are administered at Week 3. An overnight stay in the hospital is recommended for the first 24 hours. At Weeks 0, 1, 2, and 3, virology testing including HIV-1 RNA is performed with each infusion of CD4-IgG. Follow-up monitoring of patients is done once a month for 4 months for patients in Cohort II.]

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are HIV-positive.
* Are 2-12 years old and have consent of parent or legal guardian.
* Have HIV levels of 10,000 copies/ml or more on at least 2 occasions and 30 days apart (Part 2 only).
* Have been on stable, unchanged anti-HIV therapy for 3 months before study entry.

Exclusion Criteria

Children will not be eligible for this study if they:

* Have an active opportunistic (HIV-related) infection.
* Are pregnant.
* Are taking certain medications.
* Have received any vaccinations within 30 days prior to study entry.
* Have a heart problem that would affect their ability to take part in the study. (This study has been changed. The original version didn't mention heart problems.)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12
Dates: Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Shearer, Study Chair; Stuart Starr, Study Chair
Locations (8):
- United States (8):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Childrens Hosp. LA - Dept. of Ped., Div. of Clinical Immunology & Allergy, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. of Orange County, Orange, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Texas Children's Hosp. CRS, Houston, Texas

REFERENCES:
- [Background] Shearer WT, Israel RJ, Starr S, Fletcher CV, Wara D, Rathore M, Church J, DeVille J, Fenton T, Graham B, Samson P, Staprans S, McNamara J, Moye J, Maddon PJ, Olson WC. Recombinant CD4-IgG2 in human immunodeficiency virus type 1-infected children: phase 1/2 study. The Pediatric AIDS Clinical Trials Group Protocol 351 Study Team. J Infect Dis. 2000 Dec;182(6):1774-9. doi: 10.1086/317622. Epub 2000 Oct 27. PMID 11069253